CLINICAL TRIAL: NCT00793221
Title: Randomized Comparison Between Sirolimus-eluting and Everolimus-eluting Coronary Stents in Chronic Coronary Occlusions
Brief Title: Non-acute Coronary occlusIon Treated By Everolimus ELuting Stent
Acronym: CIBELES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Raul Moreno (Other)
Responsible Party: Sponsor-Investigator, Raul Moreno, Director of Invasive Cardiology, University Hospital La Paz, Madrid, Spain, Spanish Society of Cardiology
Organization: Spanish Society of Cardiology (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIBELES; HHLP003
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Artery Disease; Coronary Occlusion; Percutaneous Coronary Intervention
Keywords: Coronary stent.; Restenosis.; Coronary artery disease.; Chronic total occlusion.
MeSH Terms: conditions — Coronary Artery Disease; Coronary Occlusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus-eluting stent (Other): Implantation of sirolimus-eluting coronary stent
  Interventions: Device: Implantation of sirolimus-eluting coronary stent
- Everolimus-eluting stent (Active Comparator): Implantation of everolimus-eluting coronary stent
  Interventions: Device: Implantation of everolimus-eluting coronary stent

INTERVENTIONS:
Device: Implantation of sirolimus-eluting coronary stent — Implantation of sirolimus-eluting coronary stent after dilatation of the coronary occlusion
  Arms: Sirolimus-eluting stent
Device: Implantation of everolimus-eluting coronary stent — Implantation of everolimus-eluting coronary stent after dilatation of the coronary occlusion
  Arms: Everolimus-eluting stent

SUMMARY:
Chronic total coronary occlusions (CTO) have an especially high risk of angiographic restenosis, and need for new revascularization procedures. Drug-eluting coronary stents (DES) have demonstrated to significantly reduce the risk of restenosis and new revascularization procedures in comparison with bare-metal stents.

Most data on the efficacy of DES come from the sirolimus-eluting coronary stent Cypher (Cordis corp.), and paclitaxel-eluting coronary stent Taxus (Boston Sci.), and the Cypher stent is the only DES that has been randomly tested in CTO. Among second-generation DES, everolimus-eluting stent (EES) has shown excellent angiographic and clinical results, but this DES has not been studied in unfavourable scenario (such as CTO).

The aim of the CIBELES trial is to demonstrate the hypothesis that EES are equally effective in comparison with sirolimus-eluting stents in the treatment of CTO, in terms of angiographic efficacy considered as in-stent late lumen loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 year-old.
* A total occlusion (TIMI 0-1) with an estimated time of occlusion > 2 weeks.
* Symptomatic or silent ischaemia, or viable myocardium.
* The occlusion is suitable for percutaneous coronary intervention.
* The guidewire has crossed the occlusion, and the occlusion has been dilated with balloon or other device.

Exclusion Criteria:

* Acute myocardial infarction in the myocardial area supplied by the target vessel within 2 weeks before the inclusion in the study.
* The lesion can not be crossed with the guidewire and balloon angioplasty.
* The vessel has been previously treated percutaneously.
* The lesion is not suitable for a 2.25-3.5 coronary stent implantation.
* The patient is not willing to undergo an angiographic follow-up.
* The patient has contraindications for prolonged double (aspirin plus clopidogrel) anti-platelet therapy (e.g. allergy to aspirin, need for chronic oral anti-coagulation, or scheduled surgical intervention within 12 months.
* Pregnancy or absence of pregnancy test in women of childbearing age.
* Chronic renal failure (creatinine plasmatic values > 3.0 mg/dl).
* Plasmatic platelet count < 100.000 mm-3 or > 700.000 mm-3.
* The patient has a severe non-cardiac disease that limits his/her life expectancy to < 1 year.
* The patient is currently included in other randomized trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
In-stent late lumen loss at 9-month angiographic follow-up | 9 months

SECONDARY OUTCOMES:
Angiographic: rate of binary angiographic restenosis, rate of vessel re-occlusion, and in-segment late loss, at 9 months | 9 and 12 months
Clinical: death, myocardial infarction, new revascularization, and angina status at 1 year. | 9 and 12 months

REFERENCES:
- [Derived] Ruiz-Garcia J, Teles R, Rumoroso JR, Cyrne Carvalho H, Goicolea FJ, Moreu J, Mauri J, Mainar V, Garcia E, Moreno R; CIBELES investigators. Comparison between diabetic and non-diabetic patients after successful percutaneous coronary intervention for chronic total occlusions in the drug-eluting stent era. Rev Port Cardiol. 2015 Apr;34(4):263-70. doi: 10.1016/j.repc.2014.10.009. Epub 2015 Apr 1. PMID 25840644
- [Derived] Moreno R, Garcia E, Teles R, Rumoroso JR, Cyrne Carvalho H, Goicolea FJ, Moreu J, Mauri J, Sabate M, Mainar V, Patricio L, Valdes M, Fernandez Vazquez F, Sanchez-Recalde A, Galeote G, Jimenez-Valero S, Almeida M, Lopez de Sa E, Calvo L, Plaza I, Lopez-Sendon JL, Martin JL; CIBELES Investigators. Randomized comparison of sirolimus-eluting and everolimus-eluting coronary stents in the treatment of total coronary occlusions: results from the chronic coronary occlusion treated by everolimus-eluting stent randomized trial. Circ Cardiovasc Interv. 2013 Feb;6(1):21-8. doi: 10.1161/CIRCINTERVENTIONS.112.000076. Epub 2013 Feb 12. PMID 23403384
- [Derived] Moreno R, Garcia E, Teles RC, Almeida MS, Carvalho HC, Sabate M, Martin-Reyes R, Rumoroso JR, Galeote G, Goicolea FJ, Moreu J, Mainar V, Mauri J, Ferreira R, Valdes M, Perez de Prado A, Martin-Yuste V, Jimenez-Valero S, Sanchez-Recalde A, Calvo L, Lopez de Sa E, Macaya C, Lopez-Sendon JL. A randomised comparison between everolimus-eluting stent and sirolimus-eluting stent in chronic coronary total occlusions. Rationale and design of the CIBELES (non-acute Coronary occlusion treated by EveroLimus-Eluting Stent) trial. EuroIntervention. 2010 May;6(1):112-6. PMID 20542806